CLINICAL TRIAL: NCT00982358
Title: A 16-weeks, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Anti-inflammatory Actions of 320 mg Diovan in Patients With Type 2 Diabetes With and Without Coronary Artery Disease
Brief Title: Anti-Inflammatory Actions of Valsartan in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University of Ulm (Other)
Responsible Party: Prof. Thomas Unger, M.D., Charité-University Medicine Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489A2423; Ek#2140
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Hypertension; Type 2 Diabetes Mellitus; Coronary Artery Disease
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — Valsartan

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Valsartan (Active Comparator)
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Valsartan
  Arms: Valsartan
Other: Placebo
  Arms: Placebo

SUMMARY:
This study is designed to support the use of valsartan in the diabetic population. Two different groups will be studied, one with and one without coronary artery disease (CAD) documented by angiography.

The study is intended to demonstrate that valsartan 320 mg has an anti-inflammatory potential, reducing inflammatory serum markers as well as inflammatory gene expression, and to show that valsartan is able to improve metabolic parameters in this patient population. Furthermore, in the subgroup of patients with documented CAD this study wants to show that valsartan improves coronary perfusion.

3 Objectives

Primary objectives:

1. To demonstrate the anti-inflammatory efficacy of valsartan 160/320 mg by testing the hypothesis of superiority compared to placebo in the reduction of the inflammatory marker Tumor necrosis factor alpha (TNFα) in plasma after 16 weeks of treatment in hypertensive patients with type 2 diabetes mellitus.
2. To demonstrate the anti-inflammatory efficacy of valsartan 160/320 mg by testing the hypothesis of superiority compared to placebo in the reduction of the inflammatory marker Interleukin 6 (IL-6) in plasma after 16 weeks of treatment in hypertensive patients with type 2 diabetes mellitus.

Secondary objectives:

1. To explore the effect of 160/320 mg valsartan on parameters of insulin sensitivity.
2. To explore the effect of 160/320 mg valsartan on additional inflammatory markers in plasma [e.g. C-Reactive protein (CRP), soluble intracellular adhesion molecule-1 (sICAM-1), soluble vascular cell adhesion molecule-1 (sVCAM-1), serum amyloid A (SAA), soluble CD40 ligand (sCD40L), fibrinogen, Interleukin 1β (IL-1β), matrix metalloproteases -2, -3 and -9 (MMP-2, -3, -9), and sE-selectin)].
3. To explore the effect of 160/320 mg valsartan on inflammatory gene expression from monocytes and fat tissue.
4. To explore the effect of 160/320 mg valsartan on metabolic gene expression in fat tissue.
5. To explore the effect of 160/320 mg valsartan on coronary perfusion, in the group of patients with angiographically documented CAD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 30 and 80 years old, inclusive
* Controlled type 2 Diabetes Mellitus on stable treatment at least during the 4 weeks prior to visit 1
* Treated or untreated stage 1 (according to JNC VII Guidelines) or grade 1 (according to ESH/ESC 2003 Guidelines) hypertensive patients
* For one stratum: angiographically proven CAD
* Signed informed consent prior to any study procedure

Exclusion Criteria:

* Hypertension classified as stage 2 (or grade 2) or higher
* Normotensive patients, i.e. patients who do not have a history of high blood pressure, and who are not receiving any antihypertensive medication
* Treatment with more than 2 antihypertensive medications
* Current treatment with ARBs
* Glycated hemoglobin (HbA1c) >8.5% at Visit 1
* Current treatment with glitazones
* Myocardial infarction less than 3 months prior to Visit 1
* Total cholesterol >7.8 mmol/l
* Past diagnosis of any systemic inflammatory disease
* Known or suspected contraindications, including history of allergy to angiotensin receptor blockers
* History of hypertensive encephalopathy or cerebrovascular accident less than 1 year prior to Visit 1
* Known Keith-Wagener grade III or IV hypertensive retinopathy
* History of heart failure
* Second or third degree heart block without a pacemaker
* Concomitant unstable angina pectoris
* Concurrent potential life threatening arrhythmia or symptomatic arrhythmia
* Clinically significant valvular heart disease
* Evidence of hepatic disease as determined by any one of the following: ALT or AST values > 2 x ULN at Visit 1, a history hepatic encephalopathy, a history of esophageal varices, or a history of portocaval shunt
* Evidence of renal impairment as determined by any one of the following: serum creatinine >1.25 x ULN at visit 1, a history of dialysis, or a history of nephritic syndrome
* Sodium value <132 mmol/L at Visit 1
* Serum potassium values <3.5 mmol/L or >5.5 mmol/L at visit 1
* Any surgical or medical condition which might alter the absorption, distribution, metabolism, excretion of any drug
* Female patients who are not either post-menopausal for one year of surgically sterile, and who are not using effective contraceptive methods such as barrier method with spermicidal or an intra-uterine device. Oral contraceptive use or dermal implants as the only means of contraception are disallowed
* Pregnant or lactating females
* Any surgical or medical condition which, at the discretion of the investigator, place the patient at higher risk from his/her participation in the study, or are likely to prevent the patients from complying with the requirements of the study or completing the trial period
* History of malignancy including leukemia and lymphoma within 5 years prior to Visit 1
* History of any severe, life threatening disease within the past five years
* Any previous history of a systemic autoimmune disease
* History of drug or alcohol abuse within the last two years
* Participation in any investigational drug trial within one month prior to visit 1

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 121
Dates: Start 2004-07; Primary Completion 2006-10 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study was to evaluate the anti-inflammatory effect of VAL by analyzing the reduction of the inflammatory markers interleukin-6 (IL-6) and tumor necrosis factor alpha (TNFα) in serum after 16 weeks of treatment.

SECONDARY OUTCOMES:
To explore the effect of 160/320 mg valsartan on parameters of insulin sensitivity.
To explore the effect of 160/320 mg valsartan on additional inflammatory markers in plasma
To explore the effect of 160/320 mg valsartan on inflammatory gene expression from monocytes and fat tissue
To explore the effect of 160/320 mg valsartan on metabolic gene expression in fat tissue.
To explore the effect of 160/320 mg valsartan on coronary perfusion, in the group of patients with angiographically documented CAD

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University of Ulm, Department of Internal Medicine II, Ulm, Baden-Wurttemberg
  - Charité University Medicine Berlin, Center for Cardiovascular Research, Outpatient Clinic, Berlin, State of Berlin